CLINICAL TRIAL: NCT02661815
Title: A Phase 1b Study of Weekly Paclitaxel And Oral Ricolinostat For The Treatment Of Recurrent Platinum Resistant Ovarian, Primary Peritoneal, Or Fallopian Tube Cancer
Brief Title: A Phase 1b Study of Paclitaxel And Ricolinostat For The Treatment Of Gynecological Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decided not to move forward with further accrual.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Joyce Liu, MD, Joyce Liu, MD, MPH, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-483
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Paclitaxel; ricolinostat; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1 Expansion Cohort A (Experimental): Paclitaxel 80mg/m2 weekly days 1, 8, and 15 of a 28-day cycle Ricolinostat dosing as identified as the RP2D combination dose
  Interventions: Drug: Paclitaxel; Drug: Ricolinostat
- Phase 1 Expansion Cohort B (Experimental): Paclitaxel 70mg/m2 weekly days 1, 8, and 15 of a 28-day cycle Ricolinostat dosing as identified as the RP2D combination dose
  Interventions: Drug: Paclitaxel; Drug: Ricolinostat
- Phase 1 Expansion Cohort C (Experimental): Paclitaxel 80mg/m2 weekly days 1, 8, and 15 of a 28-day cycle Bevacizumab 10mg/kg days 1 and 15 of a 28-day cycle Ricolinostat dosing as identified as the RP2D combination dose
  Interventions: Drug: Paclitaxel; Drug: Ricolinostat; Drug: Bevacizumab
- Phase 1 Escalation Cohort (Experimental): Ricolinostat with weekly paclitaxel dosed at 80 mg/m2 per week (3 out of 4 weeks).
  Interventions: Drug: Paclitaxel; Drug: Ricolinostat

INTERVENTIONS:
Drug: Paclitaxel — Please see arm/group description.
  Other Names: Taxol
Drug: Ricolinostat — Please see arm/group description.
  Other Names: ACY-1215
Drug: Bevacizumab — Please see arm/group description.
  Other Names: Avastin
  Arms: Phase 1 Expansion Cohort C

SUMMARY:
Participants with Ovarian, Fallopian Tube, or Peritoneal Cancer that has recurred within 12 months of prior treatment that includes Platinum Chemotherapy are invited to take part in this study. This research study is studying a combination of a new chemotherapy drug called Ricolinostat together with the chemotherapy Paclitaxel and a drug called Bevacizumab as a possible treatment for this diagnosis.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies.

The FDA (the U.S. Food and Drug Administration) has not approved Ricolinostat as a treatment for any disease. The FDA has approved Paclitaxel as a treatment option for Ovarian, Fallopian Tube, or Peritoneal Cancer . The FDA has approved Bevacizumab in combination with chemotherapy as a treatment option for Ovarian, Fallopian Tube, or Peritoneal Cancer .

In this study, we are hoping to learn what is the highest dose of Ricolinostat that can be given safely together with Paclitaxel on a weekly basis or with Paclitaxel on a weekly basis and Bevacizumab every other week. Ricolinostat is a drug that stops cancer from growing by blocking the action of a protein called HDAC.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma, recurrent endometrial cancer, or recurrent cervical cancer. Histologic documentation of the original primary tumor is required via the pathology report.
* Participants must have measurable disease by RECIST 1.1 criteria. See Section 11 for the evaluation of measurable disease.
* Participants must have had at least one prior platinum-based chemotherapeutic regimen for management of primary disease (e.g., a regimen containing carboplatin, cisplatin, or another organoplatinum compound). This initial treatment may have included intraperitoneal therapy, consolidation, biologic/targeted (non-cytotoxic) agents (e.g., bevacizumab) or extended therapy administered after surgical or non-surgical assessment.

Participants are allowed to receive, but are not required to receive, biologic/targeted (non-cytotoxic) therapy as part of their primary treatment regimen.

* Participants must have recurrence within 12 months of their last platinum-containing regimen.
* Age 18 years or older
* ECOG performance status 0 or 1
* Life expectancy of greater than 16 weeks
* Participants must have normal organ and marrow function as defined below:

  * Leukocytes ≥3,000/mcL
  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Creatinine within normal institutional limits OR
  * Creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Previous toxicities from previous treatment must have resolved to grade 1 or less
* For patients in expansion cohort B, stable Grade 2 neuropathy will be allowed.
* The effects of both paclitaxel and oral ricolinostat on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participants must be able and willing to swallow pills and to absorb oral medications.
* Ability to understand and the willingness to sign a written informed consent document
* Participants must be able and willing to follow protocol instructions and schedules.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. In addition, no small molecule kinase inhibitors or any other type of investigational agent may have been administered within 4 weeks before first dose of study treatment.
* Participants may not be receiving any other investigational agents for treatment of their cancer.
* No hormonal therapy is allowed within 1 week of initiating study treatment.
* Participants may not have had radiation to >25% of the bone marrow.
* Prior treatment with a histone deacetylase inhibitor.
* Prior treatment with weekly paclitaxel for recurrent or persistent disease is not allowed. Participants may have received weekly paclitaxel as part of treatment for newly diagnosed cancer, but may not have received it as maintenance therapy following their initial therapy with platinum and taxane therapy.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to either paclitaxel or Ricolinostat. Patients who require administration of paclitaxel through a desensitization procedure are not eligible for this study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with chronic viral illnesses such as HIV-positivity and active hepatitis B or C are ineligible because they are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Any signs, symptoms, and/or radiographic evidence of a complete or partial bowel obstruction
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies as noted below, are excluded if there is any evidence of other malignancy being present within the last three years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.

  * Carcinoma in situ of the breast or cervix
  * Primary endometrial cancer meeting the following conditions: Stage not greater than IA, grade 1 or 2, no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell, or other FIGO grade 3 lesions.
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded. Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease.
* Patients with clinically significant cardiovascular disease. This includes:

  * Uncontrolled hypertension, defined as systolic greater than 140 mm Hg or diastolic greater than 90 mm Hg despite antihypertensive medications.
  * Myocardial infarction or unstable angina within 6 months prior to registration.
  * New York Heart Association (NYHA) Class II or greater congestive heart failure. (see Appendix III )
  * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or serious cardiac arrhythmia requiring medication. This does not include asymptomatic atrial fibrillation with controlled ventricular rate.
  * Any history of congenital long QT syndrome
  * The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) >500 ms within 28 days before randomization. Note: if initial QTcF is found to be > 500 ms, two additional EKGs separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is ≤500 ms, the subject meets eligibility in this regard.
* Patients with serious non-healing wound, ulcer, or bone fracture within 28 days before registration
* Patients with history of organ transplant.
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving (in contact with, invading or encasing) major vessels.
* Gastrointestinal disorders, particularly those with potential risk of perforation or fistula formation including:

  * Any of the following within 28 days of registration
  * Intra-abdominal tumor/metastases invading GI mucosa
  * Active peptic ulcer disease
  * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
  * Malabsorption syndrome.
  * Any of the following within 6 months of registration
  * Abdominal fistula
  * Gastrointestinal perforation
  * Bowel obstruction or gastric outlet obstruction
  * Note: Patients requiring drainage gastrostomy (e.g., PEG tube) and/or parenteral hydration and/or nutrition are not eligible.
  * Intraabdominal abscess.
  * Note: Complete resolution of an intraabdominal abscess must be confirmed prior to registration even if the abscess occurred more than 6 months prior to registration.
* Patients with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures which are not controlled with non-enzyme inducing anticonvulsants, any brain metastases and/or epidural disease, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months prior to the first date of study treatment.
* Major surgery within 3 months of the first dose of study drugs if there were no wound healing complications or within 6 months of the first dose of study drugs if there were wound complications.
* The following are additional exclusion criteria for patients enrolling in Expansion Cohort C:
* Uncontrolled blood pressure (>140/90). Patients should have a blood pressure of ≤140/90 taken by a medical professional within one week of starting on study
* Proteinuria >2+ on urinalysis
* Serosal involvement of the bowel that would render the patient at increased risk of gastrointestinal perforation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Liu, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massacusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were recruited in medical clinics from 03/28/2016 to 01/17/2017, the first patient was enrolled on 06/15/2016.
Period: Overall Study
Arm/Group | Phase 1 Escalation Cohort | Phase 1 Expansion Cohort A | Phase 1 Expansion Cohort B | Phase 1 Expansion Cohort C
Started | 6 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were only enrolled to the escalation cohort as the study was terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Expansion Cohort A | Phase 1 Expansion Cohort B | Phase 1 Expansion Cohort C | Phase 1 Escalation Cohort | Total
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 5 | 5
  >=65 years | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 6 | 6
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 6 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  |  | 0 | 0
  Asian |  |  |  | 1 | 1
  Native Hawaiian or Other Pacific Islander |  |  |  | 0 | 0
  Black or African American |  |  |  | 0 | 0
  White |  |  |  | 5 | 5
  More than one race |  |  |  | 0 | 0
  Unknown or Not Reported |  |  |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  |  |  | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Analysis Report on the MTD In The Dose Escalation Portion Of The Study
Description: Not assessed, the MTD was not reached as the study was terminated.
Time Frame: 2 years
Population: Data not collected as study was terminated before MTD was reached.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Escalation Cohort | Phase 1 Expansion Cohort A | Phase 1 Expansion Cohort B | Phase 1 Expansion Cohort C
Number analyzed (Participants) | 6 | 0 | 0 | 0
Participants | NA — Data not collected as study was terminated before MTD was reached |  |  |

2. Primary Outcome: Best Overall Response Measured From, Start Of Treatment To The End
Description: This is now the primary outcome measure as the study was terminated prematurely.
Time Frame: 13 months
Population: Of the six participants, four were evaluable for response by RECIST version 1.1. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least 30% decrease
Measure: Number; unit: participants
Arm/Group | Phase 1 Expansion Cohort A | Phase 1 Expansion Cohort B | Phase 1 Expansion Cohort C | Phase 1 Escalation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 4
participants
  Partial Response |  |  |  | 2
  Stable Disease |  |  |  | 2

3. Secondary Outcome: Peripheral Neurotoxicity Assessed Using TNS by Measuring 5 Categories
Description: No assessed TNS would only be assessed during escalation which we did not reach as the study was terminated.
Time Frame: 0 years
Reporting Status: Not Posted

4. Secondary Outcome: Duration Of Overall Response, Measured From The Time Measurement Criteria Are Met For PR or CR Until The First Date Recurrent Or Progressive Disease Is Objectively Documented.
Description: Not assessed, study was terminated.
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Progression-free Survival (PFS)
Description: No assessed, study was terminated.
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 1 year, 1 month.
Description: No patients were enrolled in any of the expansion cohorts.
Arm/Group | Phase 1 Expansion Cohort A | Phase 1 Expansion Cohort B | Phase 1 Expansion Cohort C | Phase 1 Escalation Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 1/6
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Expansion Cohort A (N=0) | Phase 1 Expansion Cohort B (N=0) | Phase 1 Expansion Cohort C (N=0) | Phase 1 Escalation Cohort (N=6)
syncopal episode (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Expansion Cohort A (N=0) | Phase 1 Expansion Cohort B (N=0) | Phase 1 Expansion Cohort C (N=0) | Phase 1 Escalation Cohort (N=6)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT02661815/Prot_SAP_000.pdf